CLINICAL TRIAL: NCT01812070
Title: Innovative Smartphone Application of a New Behavioral Method to Quit Smoking: Pilot Randomized Trial
Brief Title: Innovative Smartphone Application of a New Behavioral Method to Quit Smoking: Pilot Trial (Smart Quit)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7957
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Smoking
Keywords: smoking cessation; quit smoking
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Acceptance and Commitment Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT (Experimental): Acceptance & Commitment Therapy
  Interventions: Behavioral: ACT
- CBT (Active Comparator): Cognitive Behavioral Therapy
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: ACT
  Other Names: Acceptance & Commitment Therapy
  Arms: ACT
Behavioral: CBT
  Other Names: Cognitive Behavioral Therapy (CBT)
  Arms: CBT

SUMMARY:
This innovative study will compare a newly developed smartphone application for Acceptance and Commitment Therapy (ACT) to a smartphone application for traditional cognitive behavioral therapy (CBT).

DETAILED DESCRIPTION:
The study matches these National Cancer Institute (NCI) research funding priorities: (1) increasing the dissemination of smoking cessation treatments and (2) new treatment approaches to boost the effectiveness of cessation interventions.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* smokes at least five cigarettes daily for at least past 12 months
* wants to quit in the next 30 days
* interested in learning skills to quit smoking
* willing to be randomly assigned to either smartphone application
* resides in US
* has at least daily access to their own personal Apple iPhone 4, 4s, or 5
* knows how to login and download a smartphone application from Apple's "App Store" Store
* willing and able to read in English
* not participating in other smoking cessation interventions (including our other intervention studies)
* has never used the NCI's Quit Guide smartphone application.]
* willing to complete one follow-up survey
* provide email, phone, and mailing address.

Exclusion Criteria:

* The exclusion criteria are the opposite of the inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
7-day and 24-hour point prevalence quit rates | 2 months post randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- See also: Smart Quit study link — http://smartquit.org